CLINICAL TRIAL: NCT00631215
Title: Effects of Hyperbaric Oxygen Therapy on Cognitive Function on Autistic Spectrum Disordered Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pediatric Partners of Ponte Vedra (Other)
Responsible Party: Julie Buckley, MD, Pediatric Partners of Ponte Vedra
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 07.11.0005
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-01

CONDITIONS: Cognition
Keywords: Hyperbaric; Oxygen; autism
MeSH Terms: conditions — Autistic Disorder | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Healthy Adults
  Interventions: Procedure: Hyperbaric oxygen therapy

INTERVENTIONS:
Procedure: Hyperbaric oxygen therapy — Hyperbaric oxygen therapy: 1.3 atmospheres of pressure, 100%0xygen by face mask, for 60 minutes

SUMMARY:
HYPOTHESIS

1. Hyperbaric Oxygenation Therapy will be safe to use with neurotypical adults and children.
2. Hyperbaric Oxygenation Therapy will have a statistically significant positive effect on measures of cognitive function in neurotypical adults and children.
3. The improvement in cognitive function will correlate positively with the number of Hyperbaric Oxygenation Therapy sessions.
4. Treatment gains obtained from Hyperbaric Oxygenation Therapy will be maintained at follow-up, post 40 treatment sessions.

DETAILED DESCRIPTION:
Hyperbaric oxygenation chambers are FDA-approved and regulated devices. Hyperbaric oxygenation therapy (HBOT) is a medical procedure in which participants inspire enriched oxygen while their bodies are subjected to pressure greater than ambient barometric pressure at sea level (i.e., greater than 1 atmosphere absolute, or 760 mmHg). Hyperbaric oxygen therapy elevates tissue oxygen levels, thereby increasing the rate of tissue healing, and enhancing leukocyte-mediated phagocytosis. It may also elevate growth factors, which promotes angiogenesis and healing (Siddiqui, Davidson, & Mustoe, 1997).

While HBOT is most often used in wound healing and serious infections, it has been utilized in treating various disorders, most notably in cerebral palsy (Liptak, 2005; Marois & Vanasse, 2003) and other conditions, including fetal alcohol syndrome (Stoller, 2005), brain injury (Rockswold, 1993), and stroke (Helms, 2005) (see Joiner, 2002 for a review). The rationale for using HBOT in participants with neurological and developmental disorders is to relieve hypoxia, which often accompany these conditions. This leads to improvements in microcirculation and relief of cerebral edema by vasoconstriction, therefore leading to decreases in the symptom characteristics.

HBOT is implemented in various dose pressures (ATA) by practitioners for the treatment of symptoms of autism, averaging around 1.3-1.5 atmospheres for one hour sessions, for a minimum of 40 sessions. The results of HBOT are presumed to be long-term, but systematic examination of both short-term and long-term effects is currently warranted.

ELIGIBILITY:
Inclusion Criteria:

* • Males and females from 6 to 75 years of age with typical cognitive function and no neurologic or psychological diagnoses potentially impairing cognitive function

  * No anticipated changes in treatment for the study duration (e.g., diet, nutrients)

    * No additional biomedical treatments started 6 weeks prior to enrollment
    * No changes in dietary management for 3 months prior to enrollment
  * Access to Pediatric Partners on a daily basis, or as necessary for the study participation

In addition, the participant must be:

* Ambulatory or require minimum support walking
* Able to sit still for 12 minutes or longer for the purposes of test administration
* Adequate vision and hearing for the purposes of test administration, per parent
* Able to read and understand basic instructions
* Adequate arm-hand-finger coordination for computer use in outcome measurement
* Medical disorders, if present, must be stable and controlled
* Willing to participate by attending regularly scheduled appointments and completing the necessary measures
* Previous exposure to hyperbaric oxygen therapy

Exclusion Criteria:

Current otitis media Sinus infection Asthma Pulmonary cysts Emphysema Upper respiratory infection Severe claustrophobia, intolerance to being in the chamber Unstable/uncontrolled disorder of any kind

-

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-06 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
CogState touch screen measuring cognitive changes | Data will be collected according to the following schedule: prior to treatment, following 5, 15, 25, and 40 HBOT treatments, as well as at post-treatment and 1 and 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Julie Buckley, MD, Principal Investigator — President
Locations (1):
- Pediatric Partners of Ponte Vedra, Ponte Vedra Beach, Florida, United States